CLINICAL TRIAL: NCT06326593
Title: Wii Aerobic Training in Inhalation-injury Children Post-thermal Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, lectrurer of physical therapy for general surgery and dermatology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005049
Record Dates: First submitted 2024-03-14; First posted 2024-03-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Inhalation Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): Wii aerobic training (Experimental): This group included 38 children with inhalation injury post thermal burn; they will receive Wii aerobic training and conservative chest care.
  Interventions: Other: Wii aerobic training; Other: conservative chest care
- Group (B): control group (Sham Comparator): This group included 38 children with inhalation post thermal burn; they will receive conservative chest care.
  Interventions: Other: conservative chest care

INTERVENTIONS:
Other: Wii aerobic training — Nintendo Wii Fit Wii console (Nintendo Co., Ltd, Kyoto, Japan) is the main power unit of Nintendo Wii Fit. Its software includes an interactive video games that is played with a handheld, wireless remote that senses motion and requires the participant to mimic the action of their on - screen character
  Arms: Group (A): Wii aerobic training
Other: conservative chest care — Diaphragmatic deep breathing exercises Bronchial hygiene techniques Assisted cough Stretching exercises and ROM exercises for both upper and lower limbs

SUMMARY:
Inhalation injury is a composite of multiple insults including: supra glottic thermal injury, subglottic airway and alveolar poisoning, and systemic poisoning from absorbed small molecule toxins. These contaminant insults independently affect each of the pulmonary functions as well as having a direct effect on systemic physiology. Further, anatomic characteristics can predispose patients to inhalation injury. For example, an infant will develop airway obstructions much faster than an adult due to reduced airway diameter. Understanding the contributions of each of these pathologies to the patient's disease is critical to managing inhalation injury.

Wii fit aerobic training gives similar results with traditional rehabilitation practices, it causes less energy costs. This suggests that it can be a suitable rehabilitation tool for adult and elderly people with low energy levels. A review showed that video games are safe and feasible in the children with lung complications. Children' balance, aerobic and cognitive functions, quality of life improved and depressive mood decreased. WII aerobic games also make children to communicate better with other family members.

DETAILED DESCRIPTION:
This study will investigate the effects of Wii aerobic training in Inhalation-injury Children post-thermal burn. To assign patients to different treatment groups, a table of random numbers generated by a computer was used. Patients were allocated randomly into one of three groups using this method. This study will be carried out at the outpatient clinic of the faculty of physical therapy, modern university for technology and information, Om El masryeen hospital and Embaba general hosbital after referral from dermatologist. Children will perform these exercises in a room supervisor physiotherapist.

All parents of children will sign a written consent form after receiving full information about the purpose of the study, procedure, possible benefits, privacy, and use of data.

ELIGIBILITY:
Inclusion Criteria:

* Six weeks after deep second-degree thermal burn with inhalation injury (until complete healing) with 35%-40% total body surface area (TBSA), Burn size was measured using modified Lund and Browder charts.
* 12 Years to 17 Years (Child )
* Inhalation injury.
* All children suffering from retained secretions which did not respond to medical treatment.
* All children should be clinically and medically stable.
* All children should have the same medical treatment.

Exclusion Criteria:

* Children with any dysfunction that limit physical activity such as neurological disorders, chronic obstructive pulmonary disease, malignancy, cardiovascular diseases, orthopedic problems, such as fracture on the pelvic or limbs, a visual impairment, brain injury or hearing impairments and contractures.
* Children use non-invasive mechanical ventilation and intubation or need for intensive clinical support and/or transfer to the Intensive Care Unit.
* Children with other hormonal diseases

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | base line and 12 weeks.
  Forced vital capacity (FVC) will be measured by using spirometer (SP - 10 electronic hand held spirometer ) with the subject upright sitting or lying in the supine posture
forced expiratory volume in 1 second (FEV1) | base line 12 weeks
  forced expiratory volume in 1 second (FEV1) will be measured by using spirometer(SP - 10 electronic hand held spirometer) with the subject upright sitting or lying in the supine posture
peak expiratory flow (PEF) | base line 12 weeks
  peak expiratory flow (PEF) will be measured by using spirometer(SP - 10 electronic hand held spirometer ) with the subject upright sitting or lying in the supine posture

SECONDARY OUTCOMES:
Upper and lower chest expansion (2nd intercostal space, xiphoid)]) | base line 12 weeks
  chest expansion assessment
Functional capacity 6-Minute Walk Test (6-MWT) | base line 12 weeks
  that measures the maximum distance walked in a period of 6 min to assess the submaximal level of the functional capacity of the participants.
Timed Up and Go test (TUG) | base line 12 weeks
  this test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time it takes for a person to get out of the chair, walk three meters, turn around, return to the chair and sit down.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Heba Elfeky, Cairo
  - Ahmed Mohamed Ahmed Abdelhady, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferguson GD, Jelsma D, Jelsma J, Smits-Engelsman BC. The efficacy of two task-orientated interventions for children with Developmental Coordination Disorder: Neuromotor Task Training and Nintendo Wii Fit Training. Res Dev Disabil. 2013 Sep;34(9):2449-61. doi: 10.1016/j.ridd.2013.05.007. Epub 2013 Jun 7. PMID 23747936
- [Background] Mombarg R, Jelsma D, Hartman E. Effect of Wii-intervention on balance of children with poor motor performance. Res Dev Disabil. 2013 Sep;34(9):2996-3003. doi: 10.1016/j.ridd.2013.06.008. Epub 2013 Jul 2. PMID 23827983
- [Derived] Elfahl AM, Elfeky HM. Wii Aerobic Training in Inhalation-Injury Children Post-Thermal Burn: A Randomized Controlled Trial. Physiother Res Int. 2025 Apr;30(2):e70052. doi: 10.1002/pri.70052. PMID 40156880